CLINICAL TRIAL: NCT05427877
Title: Safety of Pulsing Heating Device Use on the Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Soovu Labs Inc. (Industry)
Responsible Party: Principal Investigator, Jessica Maloh, ND, Prinicipal Investigator, Integrative Skin Science and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Soovu_01
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heating Device Application (Experimental): Heating devices will be applied to the trunk and extremities of the body.
  Interventions: Device: Heating device (Heatwave Technology)

INTERVENTIONS:
Device: Heating device (Heatwave Technology) — Heating devices will be applied to the trunk and extremities of the body during the first study visit. During each heating cycle, the temperature will increase quickly from room temperature to a high of 45C and then cycle back down. Each heating cycle is 30 minutes with a 3 minute cool down period where no heat is applied. The maximum temperature used in this study is 45 degrees C (113 degrees F). There will be a total of 3 heating cycles at the visit.
  Other Names: Soovu heating devices (Heatwave Technology)

SUMMARY:
We hope to assess the safety of a recurrent heating device for pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Individuals in good general health.
* No known medical conditions that, in the investigator's opinion, may interfere with study participation.
* Subjects 18 year of age and older.

Exclusion Criteria:

* Individuals who have history of acute or chronic disease that would likely interfere with or increase the risk on study participation at the discretion of the investigator.
* Individuals with peripheral neuropathy or a neuropathic condition that would alter their ability to sense pain.
* Individuals with clinically significant unstable medical disorders that would disqualify the participant at the discretion of the investigator.
* Individuals who have history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study at the discretion of the investigator.
* Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Pain - Visual Analog Scale | 100 minutes
  Subjective reporting of pain with 10 point pain scale 0= no pain 10= very severe pain
Erythema (skin redness) | 100 minutes
  Measured with skin colorimeter
Post-inflammatory hyperpigmentation | 100 minutes
  Measured with skin colorimeter

SECONDARY OUTCOMES:
Mood and Anxiety Assessment | 100 minutes
  Survey based measure using Likert scale responses
Mood and Anxiety Assessment | 1 week
  Survey based measure using Likert scale responses
Pain - Visual Analog Scale | 1 week
  Subjective reporting of pain with 10 point pain scale 0= no pain 10= very severe pain
Erythema (skin redness) | 1 week
  Measured with skin colorimeter
Post-inflammatory hyperpigmentation | 1 week
  Measured with skin colorimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No